

## **Trial Statistical Analysis Plan**

c01837068-03

**BI Trial No.:** 1315.1

Title: A Phase I, open-label, cohort dose escalation trial with BI 836858 in

patients with refractory or relapsed acute myeloid leukemia and patients with acute myeloid leukemia in complete remission with

high risk to relapse

Including:

Protocol Amendment 1 [U11-3713-02] Protocol Amendment 2 [U11-3713-03] Protocol Amendment 3 [c02543230-04]

Investigational Product(s):

BI 836858

Responsible trial statistician(s):

Telephone:

Fax:

Date of statistical analysis plan:

09 APR 2018 REVISED

\_\_\_\_\_

**Version:** "Revised"

**** 

Proprietary confidential information

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

## 1 TABLE OF CONTENTS

| TI | TLE P | AGE | 1 |
|----|--------------|------------------------------------------------|----|
| 1 | T | ABLE OF CONTENTS | 2 |
| LI | | TABLES | |
| 2 | | IST OF ABBREVIATIONS | |
| 3 | | NTRODUCTION | |
| 4 | | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY. | |
| 5 | | | |
| | | NDPOINTS PRIMARY ENDPOINTS | |
| | 5.1<br>5.2 | SECONDARY ENDPOINTS | |
| | 5.2.1 | | |
| | 5.2.1 | | |
| | 3.2.2 | Secondary enupoints | |
| | | • | 16 |
| | | ••••• | |
| 6 | G | SENERAL ANALYSIS DEFINITIONS | 18 |
| | 6.1 | TREATMENTS | |
| | <b>6.2</b> | IMPORTANT PROTOCOL VIOLATIONS | 19 |
| | 6.3 | PATIENT SETS ANALYSED | |
| | 6.5 | POOLING OF CENTERS | |
| | 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| | 6.7 | BASELINE, TIME WINDOWS, AND CALCULATED VISITS | |
| 7 | | LANNED ANALYSES | |
| | 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| | 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| | 7.3 | TREATMENT COMPLIANCE PRIMARY ENDPOINTS | |
| | 7.4<br>7.5 | SECONDARY ENDPOINTS | |
| | 7.5.1 | Key secondary endpoint(s) | |
| | 7.5.2 | Other secondary endpoint(s) | |
| | 7.5.2 | other secondary endpoint(s) | |
| , | 7.7 | EXTENT OF EXPOSURE | |
| , | <b>7.8</b> | SAFETY ANALYSIS | |
| | <b>7.8.1</b> | Adverse events | |
| | 7.8.2 | Laboratory data | |
| | 7.8.3 | Vital signs | |
| | 7.8.4 | ECG | |
| 8 | R | EFERENCES | 33 |
| | | •••••• | 34 |
| 10 | Н | IISTORY TABLE | 35 |

# LIST OF TABLES

| able 5.2.2: 1: Derivation rules for PFS | 9 |
|---|---|
| able 5.2.2: 2: Derivation rules for TTF | 11 |
| | 13 |
| | 14 |
| able 6.1:1: Definition of analysing treatment periods | 18 |
| able 6.2: 1 Important protocol violations | 19 |
| able 7.8.1: 1: Definition of user defined AE categories (UDAEC) for Adverse Events | 27 |
| able 7.8.1: 2: User defined AE category (UDAEC) Cardiac Failure | 30 |
| able 10: 1 History table | 35 |

# 2 LIST OF ABBREVIATIONS

| Term | Definition / description |
|--------------------|----------------------------------------------------|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ATC classification | Anatomical, Therapeutic, Chemical classification |
| BI | Boehringer Ingelheim |
| BM | Bone marrow |
| BMI | Body Mass Index |
| BSA | Body Surface Area |
| BRPM | Blinded report planning meeting |
| CR | Complete Remission |
| CRi | Complete Remission with incomplete marrow recovery |
| CT | Concomitant therapy |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DBL | Data base lock |
| DILI | Drug Induced Liver Injury |
| DLT | Dose Limiting Toxicity |
| DMS | Data Management and Statistics |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic case report form |
| ЕоТ | End-of-Text |
| ICH | International Conference on Harmonisation |
| iPV | Important protocol violation |
| IRR | Infusion related reaction |
| LLQ | Lower limit of quantification |
| LVSI | Laboratory values of special interest |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQRM | Medical and Quality Review Meeting |

MTD Maximum Tolerated Dose

NE Not evaluable

PB Peripheral blood

PD Progressive disease

PFS Progression free survival

PK Pharmacokinetics

PKS Pharmacokinetic set

PR Partial remission

PT Preferred term

PV Protocol violation

REP Residual effect period

RP2D Recommended phase II dose

SAE Serious adverse event

SD Standard deviation

SDL Subject data listings

SOC System organ class

SOP Standard Operating Procedure

Treatment failure

SS Screened set

SSC Special search category

TCM Trial Clinical Monitor

TOC Table of contents

TS Treated set

TF

TSAP Trial statistical analysis plan

TTF Time to treatment failure

### 3 INTRODUCTION

As per ICH E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation. This TSAP follows the Boehringer Ingelheim (BI) internal reference (1).

This TSAP is based on the Project SAP wherever possible. Wordings like "randomisation (first administration of study treatment in non-randomised trials)" should therefore be interpreted as applicable.

SAS Version 9.2 or later version will be used for all analyses.

Version 1 of this TSAP(c01837068-02) fully specified the planned analyses for the population of patients with refractory or relapsed AML. Further enrolment of this population was stopped as of 10-JUN-2016 (for more details refer to CTP amendment 3 and the authorisation letter to continue study cohort 3 in AML patients in complete remission with high risk to relapse). In January 2018, the trial was terminated because of low patient recruitment into the CR population. This version now includes the specifications as to how the data from the CR population will be summarized a final CTR that will includes the analyses for both populations.


### 4 CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

Clarification of Residual Effect Period (REP):

According to CTP section 6.2.5, for refractory or relapsed AML patients the reporting period for adverse events is defined until 6 weeks (42 days) after last administration of study drug.

However, the residual effect period (REP) for BI 836858 is defined as 30 days. Therefore, for all safety analyses defined in this TSAP, all events occurring between first drug administration until 30 days after last drug administration will be considered on treatment. A separate table or listing will be provided with adverse events outside the on-treatment period. See TSAP section 7.8 for details.

For AML patients in CR a REP of 30 days was defined in the CTP.

For the CR patients, an abbreviated set of tables and listings will be included consisting of:

- Patient disposition
- Patient demographics
- Baseline disease characteristics
- Exposure
- Medication compliance
- Summary table of Adverse Events
- Frequency table of adverse events by highest CTCAE grade
- Frequency table of user defined adverse events by highest CTCAE grade
- Overall summary of infusion related reactions
- Listing of patients with dose related toxicities
- A frequency table of AEs by treatment, system organ class, and preferred term
- Hepatic injury (DILI)
- Listing of hepatic enzymes and bilirubin
- Summary of haemalytic laboratory values

Listings of all clinical efficacy, safety, laboratory and biomarker data will be provided.

#### 5 ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

The primary endpoints are the maximum tolerated dose (MTD) and the number of patients with of dose limiting toxicity (DLT) during the MTD evaluation period.

## Maximum tolerated dose (MTD):

MTD is defined as the highest dose studied for which the incidence of dose-limiting toxicity is no more than 17% (i.e., 1/6 patients) during the MTD evaluation period. The MTD will be defined on the basis of DLTs occurring during the MTD evaluation period of dose escalation cohorts. However, all information, including adverse events qualifying for a DLT from later times, will be considered in the final determination of the recommended Phase II dose (RP2D).

#### MTD evaluation period:

#### FOR PATIENTS WITH REFRACTORY OR RELAPSED AML,

the MTD evaluation period is defined as the time from the first administration of BI 836858 to start of the fifth administration, excluding the day of fifth administration. In case the fifth infusion will not be started, the evaluation period ends 30 days after the last administration.

#### FOR AML PATIENTS IN CR WITH HIGH RISK TO RELAPSE,

the MTD evaluation period is defined as the time from the first administration of BI 836858 to start of the third administration, excluding the day of third administration. In case the third infusion will not be started, the evaluation period ends 30 days after the last administration.

In case a patient has not completed the required number of administrations due to BI 836858 related toxicity, he/she will not be replaced and this will be considered as DLT. However, patients who have not completed the required number of administrations of BI 836858 for reasons other than BI 836858 related toxicity will be replaced.

That is, a patient will be considered evaluable for MTD assessment if he/she received at least 4 (refractory or relapsed patients) or 2 (patients in CR) administrations of BI 836858 or if he/she received less than 4 (refractory or relapsed patients) or 2 (patients in CR) administrations due to DLT.

The MTD estimate after the dose escalation part of the trial will be obtained on the basis of DLTs observed during the MTD evaluation period. However, for those patients who receive more than 4 (refractory or relapsed patients) or 2 (patients in CR) administrations of BI 836858, all AEs that constitute a DLT will be considered in the final determination of the dose recommended for Phase II.

The list of patients evaluable for MTD will be confirmed by the Trial Clinical Monitor (TCM) no later than at the last blinded report planning meeting (BRPM) before database lock (DBL) for the clinical trial report (CTR).

#### 5.2 SECONDARY ENDPOINTS

#### 5.2.1 Key secondary endpoints

Not applicable.

#### 5.2.2 Secondary endpoints

### FOR PATIENTS WITH REFRACTORY OR RELAPSED AML:

### Best overall response

The different categories possible for overall response (at a specific timepoint) are Complete remission (CR), Complete remission with incomplete blood count recovery (CRi), Partial remission (PR), Treatment failure (TF) (i.e. Resistant disease, Aplasia, Indeterminate cause, or morphologic relapse), Progressive disease (PD), and Not evaluable (NE).

Best overall response is defined as the best overall response (CR, CRi, PR, TF, PD or NE in this order) recorded since randomisation (first administration of trial medication in non-randomised trials) until the earliest of progressive disease (PD), death or last adequate disease assessment before new anti-cancer therapy.

In order to evaluate the best overall response, the investigator's assessment as given in the eCRF will be taken into account (no central review and no check versus bone marrow measurement is planned).

#### Progression free survival (PFS)

For patients with 'event' as outcome for PFS:

• PFS [days] = date of outcome - date of randomisation (date of first administration of trial medication in non-randomised trials) +1.

For patients with 'censoring' as outcome for PFS:

• PFS (censored) [days] = date of outcome - date of randomisation (date of first administration of trial medication in non-randomised trials) +1.

The censoring rules and dates of event or censoring for PFS under different scenarios are specified in Table 5.2.2:1.

Table 5.2.2: 1: Derivation rules for PFS

| Situation | Outcome (event or censored) | Date of outcome |
|---|---|---|
| Progressed according to disease assessment | event | Date of disease assessment of progression |
| Death without progression | event | Date of death |

Table 5.2.2: 1: Derivation rules for PFS (cont.)

| Situation | Outcome (event or censored) | Date of outcome |
|---|---|---|
| Alive and not progressed | censored | Date of last disease assessment |
| No disease assessment<br>performed post-baseline,<br>vital status is unknown or<br>patient is known to be alive | censored | Date of randomisation (or first treatment administration, in non-randomised trials) |
| 1 - | rapy before progression or de<br>ation and earliest of subseque | ` |
| Interval <= 7 days | event | Earliest date of disease assessment of progression or death |
| Interval > 7 days | censored | Date of last disease<br>assessment before initiation<br>of subsequent anti-cancer<br>therapy |

#### Time to treatment failure (TTF)

As some patients will receive the next line of therapy, although no formal PD may be diagnosed at the time when the next treatment is indicated, the Time to treatment failure (TTF) will be derived similarly to PFS, but will consider PD, death or start of next anti-AML therapy as events.

For patients with 'event' as outcome for TTF:

• TTF [days] = date of outcome - date of randomisation (date of first administration of trial medication in non-randomised trials) +1.

For patients with 'censoring' as outcome for TTF:

• TTF (censored) [days] = date of outcome - date of randomisation (date of first administration of trial medication in non-randomised trials) +1.

The censoring rules and dates of event or censoring for TTF under different scenarios are specified in Table 5.2.2:2.

Table 5.2.2: 2: Derivation rules for TTF

| Situation | Outcome (event or censored) | Date of outcome |
|---|---|---|
| Progressed according to disease assessment, no subsequent anti-cancer therapy | event | Date of disease assessment of progression |
| Death without progression, no subsequent anti-cancer therapy | event | Date of death |
| Subsequent anti-cancer therapy before progression or death | event | Date of first administration of subsequent anti-cancer therapy |
| Alive and not progressed,<br>no subsequent anti-cancer<br>therapy | censored | Date of last disease assessment |
| No disease assessment<br>performed post-baseline,<br>vital status is unknown or<br>patient is known to be alive,<br>no subsequent anti-cancer<br>therapy | censored | Date of randomisation (or first treatment administration, in non-randomised trials) |

## FOR AML PATIENTS IN CR WITH HIGH RISK TO RELAPSE:

Progression free survival (PFS)

Defined as for refractory/relapsed AML patients, see above.

Time to treatment failure (TTF)

Defined as for refractory/relapsed AML patients, see above.

TSAP for BI Trial No.: 1315.1 

TSAP for BI Trial No.: 1315.1 

TSAP for BI Trial No.: 1315.1 

TSAP for BI Trial No.: 1315.1 

TSAP for BI Trial No.: 1315.1 

TSAP for BI Trial No.: 1315.1 

### **6 GENERAL ANALYSIS DEFINITIONS**

#### 6.1 TREATMENTS

In this Phase I trial, treatments are not randomised (open-label, dose escalation). Different dose levels of the investigational medicinal product can arise. The data will be presented for all dose cohorts separately, in particular patients will be analysed by the treatment group initially assigned in the first treatment course.

"Analysing treatment" will be used for reporting of treatment emergent adverse events (AE) and to differentiate between screening, on-treatment, post-treatment and post-study safety data. The inequalities start date  $\leq$  onset date of AE < stop date will determine whether the AE will be assigned to the "analysing treatment" or not. <u>Table 6.1: 1</u> defines the "analysing treatment period(s)" which will be used for reporting of treatment emergent AEs and safety laboratory parameters.

Table 6.1:1: Definition of analysing treatment periods

| Analysing treatment period | Start date (including) | Stop date (excluding) |
|---|---|---|
| Screening | Date of informed consent | Date of first administration of trial medication |
| On-treatment | Date of first administration of trial medication | Start date of 'Follow-up' |
| Follow-up | Date of end of REP +1 | Start date of 'Post-study' |
| Post-study | Last date patient status obtained / last date patient known to be alive + 1 (if patient is lost to follow-up) / date of refusal + 1 day / the date patient died + 1 | During the trial: open / empty; after database lock (DBL): DBL + 1 day |
| MTD evaluation period | Date of first administration of trial medication | For patients with refractory/relapsed AML: |
| | | Date of fifth infusion or (if the fifth infusion was not administered) Date of last administration of trial medication + 30 days + 1 day |
| | | For AML patients in CR: Date of third infusion or (if the |
| | | third infusion was not<br>administered) Date of last<br>administration of trial medication +<br>30 days + 1 day |

Data recorded between the first administration of trial medication until up to 30 days (Residual effect period; REP) after the last administration of trial medication will be considered as on-treatment.

In addition, to justify the MTD determination, AEs occurring during the MTD evaluation period will be presented separately from those occurring during the complete on-treatment period.

The actual treatment codes are defined in the document entitled "5-05-o-c-treatment-setup", which can be found in the trial's DMS Section 5 within BIRDS. Labels of each analysing treatment period and analysis numbers are provided in the TSAP technical documents "ADS Plan" and "Data guide".

#### 6.2 IMPORTANT PROTOCOL VIOLATIONS

Even though no per protocol population is defined, patients with potentially important protocol violations (iPV) will be identified and documented.

Potentially important protocol violations are defined in <u>Table 6.2:1</u>. The final list of iPVs will be confirmed at the last blinded report planning meeting (BRPM) before the database lock at the time of the CTR.

Two separate iPV tables will be created for patients treated before and after the clinical hold and separately for patients with refractory/relapsed AML patients and AML patients in CR.

Table 6.2: 1 Important protocol violations

| Category/<br>Code | | Description | Comment/Example | Excluded from |
|---|---|---|---|---|
| A | | Inclusion/Exclusion Criteria | | |
| A1 | | Criteria related to safety | | |
| | A1.1 | Patient has condition that may cause additional risk from study medication | EX 7 | None |
| | A1.2 | Patient has laboratory assessments that may cause additional risk. | EX 2, EX 8-11 | None |
| | A1.3 | Patient is unable to comply with the protocol | EX 14, EX 21 | None |
| A1.4 | | Patient has condition that may interfere with evaluation of safety (and/or efficacy) | EX 3-4, EX 6, EX 12, EX 13,<br>EX15, EX 19, EX 20 | None |
| | A2 | Criteria related to efficacy | | |
| | A2.1 | Patient does not have trial diagnosis or is not part of the target population | IN 1-3, EX 1, EX 5 | None |
| В | | Legal criteria | | |

Table 6.2: 1 Important protocol violations (cont.)

| Category/ | | Description | Comment/Example | Excluded from |
|---|---|---|---|---|
| Code | | | | |
| | B1 | Informed consent not available/not done | IN 5 | All |
| | B2 | Informed consent after visit 1 | IN 5 | None |
| | В3 | Men or women who are sexually active and not using adequate contraception. | EX 16, EX 17 | None |
| | B4 | Pregnant or nursing female patient | EX 18 | None |
| | В5 | Patient's age < 18 | IN 4 | None |
| С | | Administration of trial medication not in accordance with the protocol | | |
| | C1 | Administration of trial medication not in accordance with the protocol | As marked in the eCRF, review<br>and decision at medical and<br>quality review meetings<br>(MQRM) / report planning<br>meetings (RPM) | None |
| | C2 | Continuation of treatment although criteria for re-treatment are not met | Create listing, decision at medical and quality review meetings (MQRM) / report planning meetings (RPM), see CTP section 4.1.4 | None |
| | C3 Unjustified intra-patient dose-<br>escalation | | Create listing, decision at MQRM / RPM, see CTP section 4.1.4 | None |
| | C4 | Withdrawal of patient not performed according to CTP | Create listing, decision at MQRM / RPM, see CTP section 3.3.4 | None |
| | C5 | Discontinuation of trial drug not performed according to CTP | Create listing, decision at MQRM / RPM, see CTP section 3.3.4 | None |
| D | | Restrictions | | |
| chemo-, immuno-, hormone | | Additional experimental anti-cancer, chemo-, immuno-, hormone - or radiotherapy during the study or too shortly before the study. | Create listing, decision at MQRM / RPM (section 4.2.2.1 and exclusion criteria #3, #6) | None |
| E | | Missing data | | |
| | E1 Baseline bone marrow assessment not within 14 days prior to first treatment E2 Missing disease assessment at a time point where disease assessment was required | | Create listing, decision at MQRM / RPM | None |
| | | | Create listing, decision at MQRM / RPM | None |

## 6.3 PATIENT SETS ANALYSED

- Screened set (SS): This patient set includes all patients who have signed the informed consent. The SS will be used for patient disposition tables.
- Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of trial medication. The TS will be used for all efficacy and safety analyses.

• MTD evaluable set: The MTD set consists of all patients who were entered, treated and considered evaluable for MTD determination.

The above patient sets will be defined separately for refractory/relapsed AML patients and AML patients in CR. However, due to the early enrolment stop of the refractory/relapsed AML patients, the MTD (RP2D) set is not applicable for this patient population. No combined safety analysis of both patient populations is foreseen on trial level. If deemed necessary, this will be performed on project level.

No per protocol population will be used for analyses.

#### 6.5 POOLING OF CENTERS

Not applicable because centre/country is not included in the statistical model.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

If not stated otherwise, missing data will not be imputed and remain missing. Potential outliers will be reported and analysed as observed.

Missing or incomplete AE dates are imputed according to BI standards (2).

For missing laboratory data at Visit 1 (before the very first administration of study medication) data from preceding visits will be used.

#### 6.7 BASELINE, TIME WINDOWS, AND CALCULATED VISITS

Study days and visits will be labelled according to the CTP's flow chart.

Unless otherwise specified, baseline is defined as the time-point closest to but prior to first administration of trial medication in course 1. Note that for some trial procedures (for example body weight, vital signs, laboratory tests) this may be the value measured on the same day trial medication was started. In these cases it will be assumed that the measurements were taken according to protocol, i.e. prior to first intake of any trial medication.

Laboratory values: Baseline is defined as the latest time-point before the very first administration of any trial medication in course 1. For laboratories where not only the examination date but also time are recorded, examination time has to be taken into account when defining baseline. That is, a laboratory value on the same date as the first trial drug administration is considered as baseline value if and only if the time of laboratory value is before or the same as the time of first trial drug administration.

#### 7 PLANNED ANALYSES

The labelling and display format of statistical parameters will follow the guideline "Reporting of Clinical Trials and Project Summaries" (3).

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / Standard deviation (SD) / Min / Median / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles will be preferred to mean, standard deviation, minimum and maximum.

In general, means, medians, and percentiles will be presented to one more decimal place than the raw data and SDs will be presented to two more decimal places. Minima and maxima will be presented to the same number of decimal places as the raw data.

For time-to-event analysis tables, the set of statistics is: Number of patients [N(%)], Number of patients with event [N(%)], Number of patients censored [N(%)], <Time to event> [<unit>] followed by P25 (25th percentile), median + CI, P75 (75th percentile). If not specified otherwise, the duration as well as the time to event will be displayed in months and a final decision will be made at the last RPM.

Tabulations of frequencies for categorical data will include all possible categories (even if with no count and also the missing category if there is missing data) and will display the number of observations in a category as well as the percentage (%) relative to the number of patients in the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

If a table presents only categorical data, "N (%)" will be displayed in the column header only.

Abbreviations (e.g., Wors.) or acronyms (e.g., PD) will not be displayed in tables and Subject Data Listings (SDLs) without any explanation. They will be either spelled out or explained in footnotes.

If applicable, conversion from days to weeks, months and years will be as follows:

- Weeks = days  $\div$  7
- Months =  $12 \times days \div 365.25$
- Years = days  $\div$  365.25

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Standard descriptive analyses and summary tables are planned for this section of the report. Data will be summarized by treatment group and a "total" column will be included in the summary tables.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report.

Concomitant diseases will be coded similarly as adverse events based on the most current MedDRA version. Concomitant therapies will be coded according to WHO DD. Concomitant therapies (CT) will be classified according to the Anatomical, Therapeutic, Chemical (ATC) classification system. The third ATC level will be used to categorise CTs by therapy type. In situations where a medical product may be used for more than one equally important indication, there are often several classification alternatives. As appropriate, patients receiving CTs with more than one possible ATC level-three category will be counted more than once; footnotes will clarify this possible double counting in tables.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report.

#### 7.4 PRIMARY ENDPOINTS

The primary endpoints are the MTD and the occurrence of DLT. The MTD is determined from the number of non-replaced patients with DLT during the MTD evaluation period (for the definition of MTD evaluation period refer to section 5.1).

An overall summary of patients with DLT(s) which occurred during the MTD evaluation period and the on-treatment period will be provided for each dose cohort.

Patients who were treated but replaced are not considered for the MTD determination. However, all information, including adverse events qualifying for a DLT from later times, will be considered in the final determination of the recommended Phase II dose (RP2D).

In order to describe the occurred dose escalation steps, a listing of all treated patients will be provided. This will include the initial dose of the investigational medicinal product, patient number, treatment start date, DLT in MTD evaluation period [y/n], Evaluable for MTD [y/n] and will be sorted by treatment start date.

#### 7.5 SECONDARY ENDPOINTS

### 7.5.1 Key secondary endpoint(s)

This section is not applicable as no key secondary endpoint has been specified in the protocol.

## 7.5.2 Other secondary endpoint(s)

### Best overall response:

Best overall response will be analysed descriptively. The number of treated patients and the frequency of patients by best overall response category including the corresponding percentages will be presented.

Progression-free survival (PFS) and Time to treatment failure (TTF):

PFS and TTF will be assessed based on the Kaplan-Meier method. Point estimates together with confidence intervals (based on Greenwood's method) will be provided for median PFS (if applicable). The Breslow method for handling ties will be used. The censoring rules for PFS are as stated in Section 5.2.2.

TSAP for BI Trial No.: 1315.1 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.7 EXTENT OF EXPOSURE

Standard descriptive analyses over all treatment courses will be performed. This will include a summary of the variables defined in <u>section 5.4.1</u> and will comprise a mixture of frequency and percentages, as well as summary statistics.

#### 7.8 SAFETY ANALYSIS

#### 7.8.1 Adverse events

The analyses of adverse events (AEs) will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and NOT the number of AEs.

The analyses will be based on BI standards. Adverse events will be coded with the most recent version of MedDRA. The severity of AEs will be scaled according to CTCAE version 4.03.

Reporting will be done according to version 5 of the AE guideline (6).


For analysis of AE attributes such as duration, severity, etc. multiple AE occurrence data on the CRF, will be collapsed into AE episodes provided that all of the following applies:

- The same MedDRA lowest level term was reported for the occurrences.
- The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence).
- Treatment did not change between the onset of the occurrences OR treatment changed between the onset of the occurrences, but no deterioration was observed for the later occurrence.

For each patient, all episodes with the same preferred term (PT) (system organ class, SOC) will be condensed to one AE record using a worst case approach for all AE attributes including CTCAE grading.

The analysis of adverse events will be based on the concept of treatment emergent adverse events, where a treatment emergent AE has an onset in the analyzing treatment period. All adverse events occurring before first intake of trial medication will be assigned to 'screening' and all adverse events occurring after last intake of trial medication + 30 days will be assigned to 'follow-up" (in randomised trials for listings only). For details on the treatment definition, see <a href="section 6.1">section 6.1</a>. In addition, a listing will be provided, detailing the actual treatment on the day when the adverse event started.

## Adverse events of special interest (AESIs):

Adverse events of special interest (AESIs) are defined in CTP section 5.2.2.1 as infusion related rections (IRRs) of CTCAE grade >= 3, DLTs (occurring during the MTD evaluation period or repeated treatment courses) and hepatic injury (DILI).

#### Other significant AEs:

Other significant AEs are defined as serious and non-serious AEs that lead to dose reduction or permanent discontinuation of study medication. Their incidence will be reported by severity according to CTCAE grades.

An overall summary of adverse events will be presented. This will include the number of patients with AEs by worst CTCAE grade.

The frequency of patients with adverse events will be summarised by treatment, primary system organ class and preferred term.

The system organ classes will be sorted by default alphabetically, preferred terms will be sorted by frequency (within system organ class).

AEs leading to dose reduction, AEs leading to overall permanent discontinuation, DLTs and Adverse events of special interest (AESIs) including Infusion Related Reactions (IRRs) will be tabulated.

#### Infusion related reactions (IRRs):

IRRs will be the object of special attention.

Patients with any IRR will be tabulated by treatment and worst CTCAE grade. In addition, the number of infusions and the number of IRRs will be displayed by treatment.

The duration of IRR [h] and the time since start of the respective infusion [min] together with IRR related symtoms will be tabulated by infusion number and overall.

- Duration of IRR [h] = (End time of IRR Start time of IRR) [seconds] / 3600
- Time since start of the respective infusion [min] = (Start time of IRR Start time of infusion) [seconds] / 60

The relationship between the occurrence of IRRs and infusion rate as well as the administration of premedication will be examined.

#### Fatal AEs:

AEs leading to death during the on-treatment period will be tabulated. Reported fatal AEs that occurred in the post-treatment phase will be listed.

Additionally, a table summarizing the information on deaths collected on the AE eCRF and the Patient Status eCRF will be provided.

### User defined AE categories (UDAEC):

User defined AE categories (UDAEC) for adverse events are defined in in Table 7.8.1:1. For user defined AE categories which contain sub-searches and/or two sensitivity levels (broad and narrow) all possibilities will be displayed on the UDAEC level in tables, e.g. for infusion related reactions, tables will include the UDAECs "Infusion related reactions broad" and "Infusion related reactions narrow", similarly for Bleeding: "Bleeding - SMQ Haemorrhage", "Bleeding - SMO Haemorrhage laboratory terms broad", "Bleeding - SMO Haemorrhage laboratory terms narrow", "Bleeding - SMQ Haemorrhage terms (excl. laboratory terms) narrow".

Table 7.8.1: 1: Definition of user defined AE categories (UDAEC) for Adverse Events

| Topic | UDAEC | MedDRA | (Sub-)searches | Sensitivity |
|---|---|---|---|---|
| | | code | | |
| Infusion | Infusion related | 20000021 | SMQ Anaphylactic reaction + | Narrow & |
| related | reactions | | PT Infusion related reaction <sup>1</sup> | broad |
| reactions | | | | (Algorithm) |
| Bleeding | Bleeding - SMQ | 20000040 | SMQ Haemorrhage | Narrow & |
| | Haemorrhage | | laboratory terms | broad |
| | laboratory terms | | | |
| | Bleeding - SMQ | 20000039 | SMQ Haemorrhage terms | Narrow |
| | Haemorrhage | | (excl. laboratory terms) | |
| | terms (excl. | | | |
| | laboratory terms) | | | |
| Tumor lysis | Tumor lysis | 20000219 | SMQ Tumor lysis syndrome | Narrow & |
| syndrome | syndrome | | | broad |
| | | | | (Algorithm) |

Table 7.8.1: 1: Definition of user defined AE categories (UDAEC) for Adverse Events (cont.)

| Nausea | Nausea | | BIcMQ | Narrow & broad |
|---|---|---|---|---|
| Vomiting | Vomiting | | BIcMQ | Narrow<br>&<br>broad |
| Drug related<br>hepatic<br>disorders | Drug related hepatic disorders | 20000006 | SMQ Drug related hepatic disorders <u>plus</u> the following sub-searches: | Narrow<br>&<br>broad |
| | Drug related hepatic disorders - SMQ Cholestasis and jaundice of hepatic origin | 20000009 | Cholestasis and jaundice of hepatic origin (SMQ) | Narrow<br>&<br>broad |
| | Drug related hepatic disorders -SMQ Drug related hepatic disorders - severe events only | 20000007 | Drug related hepatic disorders - severe events only (SMQ) | Narrow<br>&<br>broad |
| | Drug related hepatic disorders - SMQ Liver related investigations, signs and symptoms | 20000008 | Liver related investigations, signs and symptoms (SMQ) | Narrow<br>&<br>broad |
| | Drug related hepatic disorders - SMQ Liver- related coagulation and bleeding disturbances | 20000015 | Liver-related coagulation and bleeding disturbances (SMQ) | Narrow<br>&<br>broad |

Table 7.8.1: 1: Definition of user defined AE categories (UDAEC) for Adverse Events (cont.)

| Cardiac safety | Cardiac safety -<br>Cardiac failure<br>(tailored SMQ) <sup>2</sup> | 20000004 | Cardiac failure (tailored SMQ) <sup>2</sup> | |
|---|---|---|---|---|
| | Cardiac safety -<br>SMQ Cardiac<br>arrhythmia | 20000049 | SMQ Cardiac arrhythmia | Broad |
| | Cardiac safety -<br>SMQ Ischemia<br>heart disease | 20000043 | SMQ Ischemia heart disease | Broad |
| ALT | ALT | | BIcMQ Elevated Specific<br>Liver Function Parameters<br>sub-search1 | Narrow & broad |
| AST | AST | | BIcMQ Elevated Specific<br>Liver Function Parameters<br>sub-search2 | Narrow<br>&<br>broad |
| ALKP | ALKP | | BIcMQ Elevated Specific<br>Liver Function Parameters<br>sub-search3 | Narrow<br>&<br>broad |
| Bilirubin | Bilirubin | | BIcMQ Elevated Specific<br>Liver Function Parameters<br>sub-search5 | Narrow<br>&<br>broad |
| Neutropenia <sup>3</sup> | Neutropenia | | BIcMQ <sup>3</sup> | Broad |

<sup>&</sup>lt;sup>1</sup> The PT Infusion related reaction as collected in the eCRF will be included on both sensitivity levels (broad and narrow).

<sup>2</sup> A BIcMQ has been requested; however, as long as this is not available the terms as defined

in Table 7.8.1: 2 will be used.

<sup>&</sup>lt;sup>3</sup> Neutropenia as defined by the BIcMQ "Haematopoietic Cytopenias", Subsearch1.1.

Table 7.8.1: 2: User defined AE category (UDAEC) Cardiac Failure

| Selected PTs for Cardiac Failure |
|---------------------------------------|
| Cardiac asthma |
| Cardiac failure |
| Cardiac failure acute |
| Cardiac failure chronic |
| Cardiac failure congestive |
| Cardiac failure high output |
| Cardiac index decreased |
| Cardiac output decreased |
| Cardiogenic shock |
| Cardiomegaly |
| Cardiothoracic ratio increased |
| Dilatation ventricular |
| Left ventricular failure |
| Low cardiac output syndrome |
| Right ventricular failure |
| Oedema due to cardiac disease |
| Left ventricular dysfunction |
| Ejection fraction decreased |
| Cardiopulmonary failure |
| Diastolic dysfunction |
| Cardiac ventriculogram right abnormal |
| Cardiac ventriculogram abnormal |
| Cardiac ventriculogram left abnormal |
| Cardiac cirrhosis |
| Right ventricular dysfunction |
| Ventricular dysfunction |
| Cardiac resynchronisation therapy |
| Ventricular failure |
| Acute left ventricular failure |
| Acute right ventricular failure |
| Chronic left ventricular failure |
| Chronic right ventricular failure |
| Myocardial depression |
| Ventricular dyssynchrony |
| Systolic dysfunction |
| Neonatal cardiac failure |

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (7). The same on-treatment period as considered for the analysis of AEs will be applied for laboratory values. Patients having at least one post-baseline laboratory value will be displayed in the descriptive analyses.

Descriptive statistics, including change from baseline and frequency of patients with transitions relative to the reference range, will be provided. CTCAE grades for applicable laboratory parameters will be calculated according to CTCAE version 4.03. The following outputs will be presented:

- Worst CTCAE grade experienced during the on-treatment phase.
- Transitions of CTCAE grade from baseline to worst laboratory value, from worst to last laboratory value during the on-treatment phase, and from baseline to last laboratory value.

Patients with missing CTCAE grade at baseline or no baseline value but post baseline values will be displayed in the category "Missing CTCAE grade at baseline".

#### Possible clinically significant abnormal laboratory values:

Possible clinically significant abnormal laboratory values are defined as those laboratory values that are of CTCAE Grade  $\geq 2$  and show an increase from baseline value by at least one CTCAE grade. For those parameters for which no CTCAE has been defined, BI standard definition will be used to determine possible clinical significance. Frequency of patients with possible clinically significant abnormal laboratory values will be provided whenever applicable. If no baseline value is available but the patient has a post-baseline laboratory value of CTCAE Grade  $\geq 2$  an increase from baseline will be assumed, i.e. the laboratory value considered as possible clinically significant.

### Hepatic injury:

As defined in the CTP a hepatic injury (DILI) is defined by the following alterations of hepatic laboratory parameters:

- an elevation of AST and/or ALT >3 fold ULN combined with an elevation of total bilirubin >2 fold ULN measured in the same blood draw sample, and/or
- marked peak aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

In addition, the following definition of potential Hy's law cases was discussed with the FDA at the Pre-NDA meeting of the NSCLC submissions of the nintedanib trials 1199.13 and 1199.14 and was agreed by the authorities. Please also refer to the FDA guideline Guidance for Industry Drug- Induced Liver Injury: Premarketing Clinical Evaluation, version of July 2009.

These are defined as those cases where a combination of all of the following events occurred: any on-treatment value of ALT or AST (or both) > 3 times upper limit of normal (3 x ULN) with total bilirubin  $\ge 2$  x ULN and ALKP < 2 x ULN. The events can occur in any order, but must occur within 14 days of the previous event, i.e. the second event must occur within 14 days of the second event, etc.

All of the above combinations of elevated liver enzymes will be analysed, i.e. DILI cases as defined in the CTP and additionally the definition of potential Hy's law cases which was discussed with the FDA by the nintedanib project.

#### Handling of laboratory parameters with CTCAE grade -1:

For Uric Acid, Glomerular filtration rate (GFR) and Hypokalemia, the CTCAE grade cannot always be assigned by the laboratory parameter itself as two different CTCAE grades have the same laboratory constellation, but are distinguished by additional clinical parameter. In this case a CTCAE grade of "-1" will be assigned initially. For all analyses patients with a CTCAE grade of "-1" will be treated as

- Grade 1 for Uric Acid
- Grade 3 for GFR
- Grade 1 for Hypokalemia (Only when CTCAE version 4.03 is used)

### Handling of Urine protein (UPROZ)

With CTCAE version 4, the CTCAE grade 3 for proteinuria is defined based on 24 hrs values [g/24 hrs] only; no dipstick definition is available based on quantitative results.

High values of UPROZ (+++, ++++; labstd = 3, 4) would therefore be assigned to CTCAE grade -9, which by default is equivalent to CTCAE grade 0. To circumvent this, high values of UPROZ (+++, ++++; labstd = 3, 4) will be assigned to CTCAE grade 2.

#### 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report.

#### 7.8.4 ECG

12-lead resting ECGs are done throughout the trial and are assessed for clinically relevant results which are to be recorded as either concomitant disease or AE by the Investigator. No further ECG analysis is planned.

## **8 REFERENCES**

- 1 001-MCG-160 RD-01: "TSAP annotations", current version; IDEA for CON.
- 2 001-MCG-156\_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON.
- 3 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON.
- 4 001-MCS-36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON.
- 5 001-MCS-36-472\_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON.
- 6 001-MCG-156: "Handling and summarization of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON.
- 7 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON.

TSAP for BI Trial No.: 1315.1 

TSAP for BI Trial No.: 1315.1 

Proprietary confidential information © 2016 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10 HISTORY TABLE

Table 10: 1 History table

| Version | Date<br>(DD-Mmm-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 14-July-16 | | None | This is the final TSAP without any modification |
| Revision | 09-Apr-18 | | 4 | Added specifications for final report to include CR patients |